CLINICAL TRIAL: NCT06279520
Title: Driving Ability Evaluation System to Improve the Conditional Driving License System: Safety and Feasibility Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ja-Ho Leigh, Associate clinical professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-08-003
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Automobile Driving

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult drivers (Other): Individuals over the age of 19 who are currently driving
  Interventions: Device: VR Driving Simulator; Other: Computerized Neurocognitive Function Test; Other: Driver Test Station; Other: On-road field driving Test

INTERVENTIONS:
Device: VR Driving Simulator — Evaluation of usual road driving abilities and assessment of response capabilities in accident-prone situations through a VR driving simulator
Other: Computerized Neurocognitive Function Test — Evaluation of cognitive levels including attention and memory (the Trail Making Test, Digit Span Test, Auditory (or Visual) Continuous Performance Test , and Card Sorting)
Other: Driver Test Station — Conducting qualified tests of a person's basic physical driving ability including steering, acceleration and braking, using Driver Test Station(Autoadapt AB, Stenkullen, Sweden)
Other: On-road field driving Test — Researchers and driver's license supervisors ride in the driver's license test vehicle to evaluate the subject's actual driving ability. the validity of the VR simulator by comparing the results of the VR simulator with the actual vehicle driving ability.

SUMMARY:
The primary objective of this study is to verify the safety and validity of a VR driving simulator developed for evaluating the driving abilities in healthy adults.

This study also aims to establish indicators in VR driving simulator to evaluate high-risk group for driving, such as cognitive and physical abilities. Therefore, this study aims to measure the physical driving function and cognitive function of healthy drivers. to identify the correlation between their outcomes and the VR driving simulator's result

DETAILED DESCRIPTION:
VR driving simulator is to evaluate the driving abilities of high-risk drivers, including the elderly and those with medical conditions, potentially prone to incapacitate driving.

It aims to evaluate whether drivers who were anticipated to have impaired driving ability can handle highly risky situations for traffic accidents. The results of this study can be used to make the drivers know their status and encourage them to take safety training. Until now, the evaluation of driving abilities could only be conducted at licensing centers. However, the use of VR technology can eliminate spatial limitations, offering a promising tool for the objective assessment of driving skills.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 19 who are currently driving.
* Individuals capable of understanding and following the researcher's instructions.
* Individuals who can understand the purpose of the research and have consented to participate

Exclusion Criteria:

* Those who have not signed the consent form.
* Individuals with a history of severe dizziness or epilepsy.
* Patients with restrictions on sitting in a wheelchair or chair for more than 30 minutes.
* Patients with severe shoulder pain.
* Patients whose range of motion in major joints is restricted by more than 50%.
* Pregnant women.
* Patients with pressure sores.
* Patients with limitations on simulator use due to heterotopic ossification.
* Patients with acute fractures.
* Other patients for whom participation in the study is expected difficult.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of VR driving simulator | 2 hours
  A questionnaire evaluating symptoms of simulator sickness such as dizziness or nausea and comprehension of contents
Driving performance in simulator, measured by driving errors | 15 minutes
  Driving performance in simulator will be measured by driving errors during VR simluation of driving. These errors will be evaluated based on the criteria used for driving license tests, including violations of traffic laws.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No